CLINICAL TRIAL: NCT04999384
Title: Clinical Study Protocol AN4005X0101 An Open-Label, Multicenter, Phase 1 Study of AN4005 in Patients With Advanced Tumors
Brief Title: First in Human, Dose Escalation Study of AN4005
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adlai Nortye Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN4005X0101; AN4005 (Other: FDA)
Record Dates: First submitted 2021-07-07; First posted 2021-08-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor; Advanced Lymphoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- AN4005 dose level 0 (Active Comparator): One sentinel patient will be orally dosed at 50 mg AN4005 BID. If this dose for one cycle is deemed to be tolerable upon review of safety data and PK data, the dose of AN4005 will be escalated to next level: dose level 1.
  Interventions: Drug: AN4005-dose level 0
- AN4005 dose level 1 (Active Comparator): Three patients will be orally dosed at 100 mg AN4005 BID. Based on the number of DLT events during the first cycle, dosing decisions will be made, including add 3 patients at the same dose level (1 DLT), escalation to dose level 3 (<1/6 DLT), de-escalate to lower dose or stop (>1/6 DLT).
  Interventions: Drug: AN4005-dose level 1
- AN4005 dose level 2 (Active Comparator): Three patients will be orally dosed at 200 mg AN4005 BID. Based on the number of DLT events during the first cycle, dosing decisions will be made, including add 3 patients at the same dose level (1 DLT), escalation to dose level 3 (<1/6 DLT), de-escalate to lower dose or stop (>1/6 DLT).
  Interventions: Drug: AN4005-dose level 2
- AN4005 dose level 3 (Active Comparator): Three patients will be orally dosed at 400 mg AN4005 BID. Based on the number of DLT events during the first cycle, dosing decisions will be made, including add 3 patients at the same dose level (1 DLT), escalation to dose level 4 (<1/6 DLT), de-escalate to lower dose or stop (>1/6 DLT).
  Interventions: Drug: AN4005-dose level 3
- AN4005 dose level 4 (Active Comparator): Three patients will be orally dosed at 600 mg AN4005 BID. Based on the number of DLT events during the first cycle, dosing decisions will be made, including add 3 patients at the same dose level (1 DLT), de-escalate to lower dose or stop (>1/6 DLT).
  Interventions: Drug: AN4005-dose level 4
- AN4005 food effect (Active Comparator): The effect of a high-fat meal on the PK of AN4005 will be evaluated in a separate cohort of approximately 6 patients after a safe and clinically relevant dose is identified during the dose finding part of the study.
  Interventions: Drug: AN4005-food effect

INTERVENTIONS:
Drug: AN4005-dose level 0 — 50mg BID
  Arms: AN4005 dose level 0
Drug: AN4005-dose level 1 — 100mg BID
  Arms: AN4005 dose level 1
Drug: AN4005-dose level 2 — 200mg BID
  Arms: AN4005 dose level 2
Drug: AN4005-dose level 3 — 400mg BID
  Arms: AN4005 dose level 3
Drug: AN4005-dose level 4 — 600mg BID
  Arms: AN4005 dose level 4
Drug: AN4005-food effect — Dose to be determined upon the MTD determination
  Arms: AN4005 food effect

SUMMARY:
Open-label, multicenter, phase 1 study to investigate the safety, tolerability, and PK of AN4005 in patients with advanced tumors. This study is a first-in-human, dose escalation study with the objective to establish the MTD and/or RP2D of AN4005.

Except for Dose Level 0 (50 mg), a traditional "3 + 3 design" will be utilized for dose finding with dose escalation and/or de-escalation as appropriate.

DETAILED DESCRIPTION:
In this study, one sentinel patient will be dosed at 50 mg first, then increasing doses of AN4005 will be administered to cohorts of 3 subjects, at doses ranging from 100 mg twice daily (BID) to 600 mg BID (see the table below). The proposed starting dose, 50 mg BID, has been selected based on integrated data from nonclinical studies. If 50 mg BID for one cycle is deemed to be tolerable upon review of safety data, the dose of AN4005 will be escalated to 100 mg BID in a cohort of 3 patients, and further dose escalations will be performed in separate cohorts based on review of data from all preceding cohorts. The dose escalation will be conducted in a sequential manner. Intermediate dose levels (decrement) may be explored. Decisions with regard to dose escalation to next dose level will be made jointly by the investigators and the sponsor. AE data collected for approximately 90 days following the end of exposure will also be used to inform the final dose and schedule. A minimum of 6 patients will be treated at the MTD/RP2D.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years at the time of informed consent and have provided signed informed consent for the trial.

  2. Willing and able to comply with all aspects of the protocol.

  3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

  4. Life expectancy ≥ 3 months.

  5. Subjects with histologically or cytologically confirmed advanced solid tumors that are metastatic or unresectable, or relapsed or refractory (r/r) lymphoma, and for whom standard life-prolonging measures are not available. Types of lymphoma may include, but are not limited to, natural killer (NK)/T-cell lymphoma, classic Hodgkin lymphoma (cHL), peripheral T-cell lymphoma (PTCL), and diffuse large B-cell lymphoma (DLBCL).

  6. No standard therapy available or standard therapy is considered unsuitable or intolerable according to the Investigator.

  7. Patients with or without measurable disease are considered eligible. Patients who have measurable disease as assessed by the local site investigator and/or radiologist. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

  8. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. If previously treated with anti-PD-1/PD-L1 therapy, tumor tissue sample obtained following the most recent anti-PD-1/PD-L1 therapy is required. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue. For patients with specific types of lymphomas, bone marrow biopsy will be required as appropriate.

  9. Left ventricular ejection fraction (LVEF) greater than 50% on echocardiography or multiple gated acquisition (MUGA) scan.

  10. Patient has organ function as shown by the following:
  1. Absolute neutrophil count (ANC) ≥1.5 x 109/L.
  2. Hemoglobin ≥8 g/dL (which may be reached by transfusion).
  3. Platelets ≥100 x 109/L (which may be reached by transfusion).
  4. International normalized ratio (INR) ≤1.5.
  5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 x upper limit of normal (ULN) or <5.0 x ULN if liver metastases are present.
  6. Total serum bilirubin ≤ ULN or ≤1.5 x ULN if liver metastases are present; or total bilirubin ≤3.0 x ULN with direct bilirubin below or within normal range in patients with well documented Gilbert's Syndrome. Gilbert's syndrome is defined as presence of episodes of unconjugated hyperbilirubinemia with normal results from cells blood count (including normal reticulocyte count and blood smear), normal liver function test results, and absence of other contributing disease processes at the time of diagnosis.
  7. Creatinine clearance (CrCL) >60 mL/min calculated by the Cockcroft-Gault Equation.

     11. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  <!-- -->

  1. Not a woman of childbearing potential Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks prior to Screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment, is she considered not of child-bearing potential.
  2. Woman of childbearing potential who agrees to follow contraceptive guidance during the treatment period and for at least 90 days after the last dose of study treatment.

Highly effective contraception is defined as either:

* Total abstinence: When this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Female sterilization: When the female study patient has had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
* Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female study patients, the vasectomized male partner should be the sole partner for that patient.
* Using a combination of any two of the following:

  * Placement of an intrauterine device (IUD) or intrauterine system (IUS), and
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
  * Hormonal contraception methods (e.g., oral, injected, implanted).

    12. A male participant must agree to use contraception during the treatment period and for at least 90 days after the last dose of the study treatment.

Exclusion Criteria:

1. Have been discontinued treatment due to a Grade 3 or higher immune-related AE (irAE) from prior anti-PD-1or anti-PD-L1 therapy, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
2. Have received prior systemic anti-cancer therapy including investigational oncology agents within 4 weeks or 5 half-lives, whichever is shorter.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or returned to baseline. Participants with ≤ Grade 2 neuropathy or alopecia may be eligible.
3. At least 6 weeks must have elapsed since CAR-T infusion and subjects must have experienced disease progression, and not have residual circulating CAR-T cells in peripheral blood (based on local assessment). Any encountered treatment-related toxicities must have resolved to Grade ≤1.
4. Have received prior palliative radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
5. Uncontrolled tumor-related pain.
6. Have received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Non live COVID vaccinations or boosters should not occur within 30 days prior to the first dose of study drug and during Cycle 1.
7. Are currently participating in a study of an investigational agent or investigational device within 4 weeks or less than 5 half-lives, prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been at least 4 weeks after the last dose of the previous investigational agent (see Number 2 above).
8. Have had an allogenic tissue (e.g., bone marrow or stem cells)/solid organ transplant within the past 5 years.
9. Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
10. With a history of another primary malignancy within the past 2 years, with the following exceptions: basal or squamous cell skin cancer, or carcinoma in situ of the cervix or breast that has undergone potentially curative therapy; or patients with a prior history of or clinically stable concurrent malignancy provided the malignancy is clinically insignificant, no treatment is required, and the patient is clinically stable.
11. Have known severe hypersensitivity to study treatment components.
12. Have an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
13. Have a history of (non-infectious) pneumonitis that has required steroids or have current pneumonitis.
14. Have an active infection requiring systemic therapy within 2 weeks prior to the first dose of the study drug.
15. Significant cardiovascular (CV) impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of the study drug; or cardiac arrhythmia requiring medical treatment (including oral anticoagulation). Patients who meet the following criteria should be excluded: a) A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >470 milliseconds (ms) using Fredericia's QT correction formula). b) A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome). c) The use of concomitant medications that prolong the QT/QTc interval.
16. Major surgery within 4 weeks before the first dose of the study drug. Note: If participant received major surgery, they must have recovered adequately from surgery and the toxicity and/or complications requiring the intervention prior to starting study treatment.
17. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the oral bioavailability of the investigational drugs.
18. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
19. Have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study, e.g. history of or active major depressive episode, bipolar disorder, obsessive-compulsive disorder, schizophrenia, or history of suicidal attempt or ideation, homicidal ideation (e.g., risk of doing harm to self or others), or patients with active severe personality disorders (defined according to Diagnostic and Statistical Manual of Mental Disorders [DSM V]) are not eligible. Note: For patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous six weeks prior to start of study drug.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 90 days after the last dose of study treatment.
21. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures >/=1 time per month.
22. Leptomeningeal disease.
23. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated but without evidence that disease has been clinically stable for >/=2 weeks prior to the first dose of the study drug.
24. Oral or IV antibiotics within 2 weeks prior to the first dose of the study drug (except for prophylactic dose).
25. Active tuberculosis.
26. Patient is currently being treated with drugs known to be strong cytochromes P450 (CYP)3A4, inhibitors or inducers; UGT inducers or inhibitors; inhibitors of P-gP; sensitive substrates for CPY3A4, CYP2C9, CPY2C19 or P-gP (Appendix 4: List of Concomitant Drugs to Avoid Two Weeks Prior to and During Patient Enrollment) and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
27. Patient has a history of non-compliance to any medical regimen or inability to grant consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with any adverse events (AEs), serious adverse events (SAEs), withdrawal due to AEs, dose interruptions and reductions | Up to approximately 1 year
  All AEs, SAEs and dose modifications will be collected
Number of participants with dose limiting toxicities (DLTs) | Up to 28 days
  An event is considered to be a DLT if the event occurs within the first 28 days of treatment and meets the dose-limiting toxicity criteria, unless it can be clearly established that the event is unrelated to treatment
Number of participants with clinically significant changes in laboratory parameters, vital signs, physical examination and organ-specific parameters | Up to approximately 1 year
  Blood and urine samples will be collected for analysis of lab parameters. Vital signs, physical examinations and organ-specific parameters will be collected at specified time points

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of AN4005 | Baseline and up to approximately 1 year
  Blood samples will be collected at given time points to determine the Cmax of AN4005
Area under the plasma concentration-time curve (AUC) extrapolated from time zero to infinity (AUC[0-inf]) of AN4005 | Up to approximately 1 year
  Blood samples will be collected at given time points to determine the AUC (0-inf) of AN4005
AUC from time zero to the last quantifiable concentration after dosing (AUC[0-t]) of AN4005 | Up to approximately 1 year
  Blood samples will be collected at given time points to determine the AUC (0-t) of AN4005
AUC over the dosing interval tau (AUC[0-tau]) of AN4005 | Up to approximately 1 year
  Blood samples will be collected at given time points to determine the AUC (0-tau) of AN4005
Terminal phase half-life (t1/2) of AN4005 | Up to approximately 1 year
  Blood samples will be collected at given time points to determine the half-life of AN4005
Oral clearance (CL/F) of AN4005 | Up to approximately 1 year
  Blood samples will be collected at given time points to determine the CL/F of AN4005
Accumulation ratio (AR) of AN4005 | Up to approximately 1 year
  Blood samples will be collected at given time points to determine the AR of AN4005
Participants with solid tumors: Overall response rate (ORR) based on Evaluation Criteria In Solid Tumors (RECIST) 1.1 | Up to approximately 1 year
  ORR is defined as the percentage of participants achieving a confirmed complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. All solid tumor cohorts will score ORR by investigator assessment
Participants with lymphoma: ORR based on Lugano criteria | Up to approximately 1 year
  ORR is defined as the percentage of participants achieving CR or PR based on Lugano criteria
Evaluate progression free survival (PFS) of participants | Up to approximately 1 year
  PFS is defined as the time of participants free from first dose of treatment until radiographic progression based on RECIST 1.1 or Lugano criteria or death due to any cause, whichever is earlier. Median PFS will be estimated using the Kaplan-Meier product limit method and provided graphically
Evaluate disease control rate (DCR) of participants | Up to approximately 1 year
  DCR is defined as the proportion of patients with a BOR of CR, PR or stable disease (SD) by investigator review
Evaluate duration of Response (DOR) of participants | Up to approximately 1 year
  DOR is defined as the time from first evidence of response (CR or PR per RECIST 1.1) to earlier date of disease progression or death due to any cause, as determined by ICR
Evaluate complete remission rate (CRR) of participants | Up to approximately 1 year
  CRR is defined as the proportion of patients with a best overall response of CR by investigator review. For Lugano 2014 Criteria for lymphomas, CR is defined as disappearance of all clinical/radiographic evidence of disease, regression of lymph nodes to normal size, absence of spleen, liver, and bone marrow involvement
Evaluate overall survival (OS) of participants | Up to approximately 1 year
  OS is defined as the time from first dose of AN4005 until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Dryer, Study Director — Adlai Nortye USA Inc
Locations (7):
- United States (4):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Montefiore Einstein Cancer Center, The Bronx, New York
  - Prisma Health Institute for Translational Oncology Research, Greenville, South Carolina
  - Next Virginia, Fairfax, Virginia
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No